CLINICAL TRIAL: NCT04223960
Title: A First-in-human, Randomized, Double-blinded, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Bioavailability and Food-effects of EA1080 in Healthy Caucasian and Japanese Male Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Bioavailability, and Food-effects of EA1080 in Healthy Caucasian and Japanese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: EA1080-CP1; 2019-001886-34 (EudraCT Number)
Record Dates: First submitted 2020-01-02; First posted 2020-01-13 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
Keywords: EA1080; Pharmacokinetics; Food effect study; Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (26):
- Part A: SAD, EA1080 Formulation A in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation A or matching placebo orally, once on Day 1 of SAD part of the study. In SAD, there will be a maximum of 7 dose levels (three-four planned cohorts and three optional cohorts).
  Interventions: Drug: EA1080; Drug: EA1080-matching placebo
- Part A: SAD, EA1080 Formulation B in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation B or matching placebo orally, once on Day 1 of SAD part of the study. In SAD, there will be a maximum of 7 dose levels (three-four planned cohorts and three optional cohorts).
  Interventions: Drug: EA1080; Drug: EA1080-matching placebo
- Part A: SAD, EA1080 Formulation C in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation C or matching placebo orally, once on Day 1 of SAD part of the study. In SAD, there will be a maximum of 7 dose levels (three-four planned cohorts and three optional cohorts).
  Interventions: Drug: EA1080; Drug: EA1080-matching placebo
- Part A: SAD, EA1080 Formulation D in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation D or matching placebo orally, once on Day 1 of SAD part of the study. In SAD, there will be a maximum of 7 dose levels (three-four planned cohorts and three optional cohorts).
  Interventions: Drug: EA1080; Drug: EA1080-matching placebo
- Part A: SAD, EA1080 in Healthy Japanese Participants (Optional) (Experimental): Healthy Japanese participants will receive any EA1080 formulation (Formulation A, Formulation B, Formulation C, and Formulation D) or matching placebo orally, once on Day 1 of SAD part of the study. There will be a maximum of six dose levels (three planned and three optional cohorts) per formulation.
  Interventions: Drug: EA1080; Drug: EA1080-matching placebo
- Part A: FE and Optional BA in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 on Day 1 and Day 8 in selected formulations (Formulation A, Formulation B, Formulation C, and Formulation D) in fed and fasted states. These formulations may be tested in any order or combination up to eight- way crossover design. The order will be dependent on the treatment sequence in which participants will be allocated to treatment. A washout period of 7 days will be maintained between the dosing days of each treatment periods.
  Interventions: Drug: EA1080
- Part A: FE and Optional BA, in Healthy Japanese Participants (Experimental): Healthy Japanese participants will receive EA1080 on Day 1 and Day 8 in selected formulations (Formulation A, Formulation B, Formulation C, and Formulation D) in fed and fasted states. These formulations may be tested in any order or combination up to four-way crossover design. The order will be dependent on the treatment sequence in which participants will be allocated to treatment. A washout period of 7 days will be maintained between the dosing days of each treatment periods.
  Interventions: Drug: EA1080
- Part A: MAD, EA1080 Formulation A in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation A or matching placebo orally, once on Day 1 then multiple daily doses beginning on Day 8 up to Day 21 in MAD part of the study. In MAD, there will be a maximum of 6 dose levels (three planned cohorts and three optional cohorts).
  Interventions: Drug: EA1080; Drug: EA1080-matching placebo
- Part A: MAD, EA1080 Formulation B in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation B or matching placebo orally, once on Day 1 then multiple daily doses beginning on Day 8 up to Day 21 in MAD part of the study. In MAD, there will be a maximum of 6 dose levels (three planned cohorts and three optional cohorts).
  Interventions: Drug: EA1080; Drug: EA1080-matching placebo
- Part A: MAD, EA1080 Formulation C in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation C or matching placebo orally, once on Day 1 then multiple daily doses beginning on Day 8 up to Day 21 in MAD part of the study. In MAD, there will be a maximum of 6 dose levels (three planned cohorts and three optional cohorts).
  Interventions: Drug: EA1080; Drug: EA1080-matching placebo
- Part A: MAD, EA1080 Formulation D in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation D or matching placebo orally, once on Day 1 then multiple daily doses beginning on Day 8 up to Day 21 in MAD part of the study. In MAD, there will be a maximum of 6 dose levels (three planned dose level and three optional).
  Interventions: Drug: EA1080; Drug: EA1080-matching placebo
- Part A: MAD, EA1080 in Healthy Japanese Participants (Optional) (Experimental): Healthy Japanese participants will receive any EA1080 formulation (Formulation A, Formulation B, Formulation C, and Formulation D) or matching placebo orally, once on Day 1 then multiple daily doses beginning on Day 8 up to Day 21 in MAD part of the study. In MAD, there will be a maximum of 6 dose levels (three planned dose level and three optional) per formulation.
  Interventions: Drug: EA1080; Drug: EA1080-matching placebo
- Part B: SAD, EA1080 Formulation E in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation E or matching placebo orally, once on Day 1 of SAD part of the study (three planned cohorts and six optional cohorts).
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: SAD, EA1080 Formulation E in Healthy Japanese Participants (Experimental): Healthy Japanese participants will receive EA1080 Formulation E or matching placebo orally, once on Day 1 of SAD part of the study (three planned cohorts and six optional cohorts).
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: SAD, EA1080 Formulation F in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation F or matching placebo orally, once on Day 1 of SAD part of the study (three planned cohorts and six optional cohorts).
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: SAD, EA1080 Formulation F in Healthy Japanese Participants (Experimental): Healthy Japanese participants will receive EA1080 Formulation E or matching placebo orally, once on Day 1 of SAD part of the study (three planned cohorts and six optional cohorts).
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: SAD-FE, EA1080 Formulation E in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation E or matching placebo on Day 1 in fasted state followed by EA1080 Formulation E on Day 8 in fed states. A washout period of 6 days will be maintained between the dosing days.
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: SAD-FE, EA1080 Formulation E in Healthy Japanese Participants (Experimental): Healthy Japanese participants will receive EA1080 Formulation E or matching placebo on Day 1 in fasted state followed by EA1080 Formulation E on Day 8 in fed states. A washout period of 6 days will be maintained between the dosing days.
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: SAD-FE, EA1080 Formulation F in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation F or matching placebo on Day 1 in fasted state followed by EA1080 Formulation F on Day 8 in fed states. A washout period of 6 days will be maintained between the dosing days.
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: SAD-FE, EA1080 Formulation F in Healthy Japanese Participants (Experimental): Healthy Japanese participants will receive EA1080 Formulation F or matching placebo on Day 1 in fasted state followed by EA1080 Formulation F on Day 8 in fed states. A washout period of 6 days will be maintained between the dosing days.
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: FE/BA, in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 on Days 1 8 and 15 in selected formulations (Formulation E in fasted state, Formulation F in fasted state, Formulation F in fed state). These formulations will be tested in a crossover design. The order will be dependent on the treatment sequence in which participants will be allocated to treatment. A washout period of 6 days will be maintained between the dosing days of each treatment periods.
  Interventions: Drug: EA1080
- Part B: FE/BA, in Healthy Japanese Participants (Experimental): Healthy Japanese participants will receive EA1080 on Days 1 8 and 15 in selected formulations (Formulation E in fasted state, Formulation F in fasted state, Formulation F in fed state). These formulations will be tested in a crossover design. The order will be dependent on the treatment sequence in which participants will be allocated to treatment. A washout period of 6 days will be maintained between the dosing days of each treatment periods.
  Interventions: Drug: EA1080
- Part B: MAD, EA1080 Formulation E in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation E or matching placebo orally, once on Day 1 then multiple daily doses beginning on Day 8 up to Day 17 in Part B, MAD of the study. In Part B, MAD, there will be a maximum of 6 dose levels (one-three planned dose level and six optional).
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: MAD, EA1080 Formulation E in Healthy Japanese Participants (Experimental): Healthy Japanese participants will receive EA1080 Formulation E or matching placebo orally, once on Day 1 then multiple daily doses beginning on Day 8 up to Day 17 in Part B, MAD of the study. In Part B, MAD, there will be a maximum of 6 dose levels (one-three planned dose level and six optional).
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: MAD, EA1080 Formulation F in Healthy Caucasian Participants (Experimental): Healthy Caucasian participants will receive EA1080 Formulation F or matching placebo orally, once on Day 1 then multiple daily doses beginning on Day 8 up to Day 17 in Part B, MAD of the study. In Part B, MAD, there will be a maximum of 6 dose levels (one-three planned dose level and six optional).
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080
- Part B: MAD, EA1080 Formulation F in Healthy Japanese Participants (Experimental): Healthy Japanese participants will receive EA1080 Formulation F or matching placebo orally, once on Day 1 then multiple daily doses beginning on Day 8 up to Day 17 in Part B, MAD of the study. In Part B, MAD, there will be a maximum of 6 dose levels (one-three planned dose level and six optional).
  Interventions: Drug: EA1080-matching placebo; Drug: EA1080

INTERVENTIONS:
Drug: EA1080 — EA1080 Formulation A.
  Arms: Part A: FE and Optional BA in Healthy Caucasian Participants; Part A: FE and Optional BA, in Healthy Japanese Participants; Part A: MAD, EA1080 Formulation A in Healthy Caucasian Participants; Part A: MAD, EA1080 in Healthy Japanese Participants (Optional); Part A: SAD, EA1080 Formulation A in Healthy Caucasian Participants; Part A: SAD, EA1080 in Healthy Japanese Participants (Optional)
Drug: EA1080 — EA1080 Formulation B.
  Arms: Part A: FE and Optional BA in Healthy Caucasian Participants; Part A: FE and Optional BA, in Healthy Japanese Participants; Part A: MAD, EA1080 Formulation B in Healthy Caucasian Participants; Part A: MAD, EA1080 in Healthy Japanese Participants (Optional); Part A: SAD, EA1080 Formulation B in Healthy Caucasian Participants; Part A: SAD, EA1080 in Healthy Japanese Participants (Optional)
Drug: EA1080 — EA1080 Formulation C.
  Arms: Part A: FE and Optional BA in Healthy Caucasian Participants; Part A: FE and Optional BA, in Healthy Japanese Participants; Part A: MAD, EA1080 Formulation C in Healthy Caucasian Participants; Part A: MAD, EA1080 in Healthy Japanese Participants (Optional); Part A: SAD, EA1080 Formulation C in Healthy Caucasian Participants; Part A: SAD, EA1080 in Healthy Japanese Participants (Optional)
Drug: EA1080 — EA1080 Formulation D.
  Arms: Part A: FE and Optional BA in Healthy Caucasian Participants; Part A: FE and Optional BA, in Healthy Japanese Participants; Part A: MAD, EA1080 Formulation D in Healthy Caucasian Participants; Part A: MAD, EA1080 in Healthy Japanese Participants (Optional); Part A: SAD, EA1080 Formulation D in Healthy Caucasian Participants; Part A: SAD, EA1080 in Healthy Japanese Participants (Optional)
Drug: EA1080-matching placebo — EA1080-matching placebo.
  Arms: Part A: MAD, EA1080 Formulation A in Healthy Caucasian Participants; Part A: MAD, EA1080 Formulation B in Healthy Caucasian Participants; Part A: MAD, EA1080 Formulation C in Healthy Caucasian Participants; Part A: MAD, EA1080 Formulation D in Healthy Caucasian Participants; Part A: MAD, EA1080 in Healthy Japanese Participants (Optional); Part A: SAD, EA1080 Formulation A in Healthy Caucasian Participants; Part A: SAD, EA1080 Formulation B in Healthy Caucasian Participants; Part A: SAD, EA1080 Formulation C in Healthy Caucasian Participants; Part A: SAD, EA1080 Formulation D in Healthy Caucasian Participants; Part A: SAD, EA1080 in Healthy Japanese Participants (Optional); Part B: MAD, EA1080 Formulation E in Healthy Caucasian Participants; Part B: MAD, EA1080 Formulation E in Healthy Japanese Participants; Part B: MAD, EA1080 Formulation F in Healthy Caucasian Participants; Part B: MAD, EA1080 Formulation F in Healthy Japanese Participants; Part B: SAD, EA1080 Formulation E in Healthy Caucasian Participants; Part B: SAD, EA1080 Formulation E in Healthy Japanese Participants; Part B: SAD, EA1080 Formulation F in Healthy Caucasian Participants; Part B: SAD, EA1080 Formulation F in Healthy Japanese Participants; Part B: SAD-FE, EA1080 Formulation E in Healthy Caucasian Participants; Part B: SAD-FE, EA1080 Formulation E in Healthy Japanese Participants; Part B: SAD-FE, EA1080 Formulation F in Healthy Caucasian Participants; Part B: SAD-FE, EA1080 Formulation F in Healthy Japanese Participants
Drug: EA1080 — EA1080 Formulation E.
  Arms: Part B: FE/BA, in Healthy Caucasian Participants; Part B: FE/BA, in Healthy Japanese Participants; Part B: MAD, EA1080 Formulation E in Healthy Caucasian Participants; Part B: MAD, EA1080 Formulation E in Healthy Japanese Participants; Part B: SAD, EA1080 Formulation E in Healthy Caucasian Participants; Part B: SAD, EA1080 Formulation E in Healthy Japanese Participants; Part B: SAD-FE, EA1080 Formulation E in Healthy Caucasian Participants; Part B: SAD-FE, EA1080 Formulation E in Healthy Japanese Participants
Drug: EA1080 — EA1080 Formulation F.
  Arms: Part B: FE/BA, in Healthy Caucasian Participants; Part B: FE/BA, in Healthy Japanese Participants; Part B: MAD, EA1080 Formulation F in Healthy Caucasian Participants; Part B: MAD, EA1080 Formulation F in Healthy Japanese Participants; Part B: SAD, EA1080 Formulation F in Healthy Caucasian Participants; Part B: SAD, EA1080 Formulation F in Healthy Japanese Participants; Part B: SAD-FE, EA1080 Formulation F in Healthy Caucasian Participants; Part B: SAD-FE, EA1080 Formulation F in Healthy Japanese Participants

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of EA1080 following single and multiple ascending oral doses in healthy Caucasian and Japanese male participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called EA1080. EA1080 is being tested to find a safe and well-tolerated dose in healthy Caucasian and Japanese male participants. The study consists of 2 parts as mentioned below:

Part A: This part of the study is fully adaptive and will be performed in three sub-parts as follows:

* Single ascending dose (SAD)
* Food Effect (FE) and optional bioavailability
* Multiple ascending dose (MAD)

Part B: This part of study is comprised of four sub-parts to assess Formulation E and Formulation F as follows:

* SAD
* An additional FE period in SAD cohorts (SAD-FE)
* Food Effect and bioavailability (FE/BA)
* MAD

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for enrolment in this study:

1. Participants in Caucasian cohorts must be healthy males, aged greater than or equal (>=) 18 to less than or equal to (<=) 45 years at the date of signing informed consent
2. Participants in Japanese cohorts must be healthy males, aged >=20 to <=45 years at the date of signing informed consent
3. Participants must have a body mass index (BMI) between 18.5-25.0 kilogram per square meter (kg/m^2) inclusive at screening, Day -3, Day -2 or Day -1.

Exclusion Criteria:

Participants will be excluded from enrolment in this study if they meet any of the following criteria:

1. Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening
2. Consumption of herbal remedies or dietary supplements containing St. John's Wort 30 days before the first day of dosing
3. Has donated or lost 400 milliliter (mL) blood or more within the last 16 weeks preceding the first day of dosing
4. An inability to follow a standardised diet and meal schedule or inability to fast, as required during the study
5. Prior screen failure (where the cause of the screen failure is not deemed to be temporary), randomisation, participation, or enrolment in this study. Participants who initially failed due to temporary non-medically significant issues are eligible for re-screening once the cause has resolved
6. Participants with veins on either arm that are unsuitable for intravenous puncture or cannulation (example, veins that are difficult to locate, or a tendency to rupture during puncture)
7. Participants with any medical condition which may cause raised intracranial pressure, participants with new or changing headaches, and participants with history of head or spinal trauma
8. An absolute lymphocyte count below 0.9*10^9 per liter (/L) at screening or on Day -1
9. Participants in receipt of any vaccination for Corona virus disease (COVID-19) within 14 days prior to the first dose administration.
10. History of COVID-19 polymerase chain reaction (PCR) positivity within 3 months of Day 1, suspected COVID-19 based on clinical presentation within 3 months of Day 1, or presence of clinically relevant long term sequelae of COVID-19.
11. Unwillingness to receive COVID-19 testing per local or site COVID-19 guidance.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 184 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2023-08-06 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to approximately 3 year 4 months
Parts A and B: Percentage of Participants With Clinically Significant Change From Baseline in Laboratory Parameter Values | Up to approximately 3 year 4 months
Parts A and B: Percentage of Participants With Abnormal, Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Findings | Up to approximately 3 year 4 months
Parts A and B: Percentage of Participants With Clinically Significant Change From Baseline in Vital Sign Values | Up to approximately 3 year 4 months

SECONDARY OUTCOMES:
Parts A and B: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) of EA1080 and its Metabolite | Part A and B, SAD: Pre-dose (Day 1) and up to Day 8; Part A, FE and Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22; MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and B: T1/2: Terminal Half-life of EA1080 and its Metabolite | Part A and B, SAD: Pre-dose (Day 1) and up to Day 8; Part A, FE and Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22; MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and B: Cmax: Maximum Observed Plasma Concentration of EA1080 and its Metabolite | Part A and B, SAD: Pre-dose (Day 1) and up to Day 8; Part A, FE and Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22; MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and B: AUC (0-t): Area Under the Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration of EA1080 and its Metabolite | Part A and B, SAD: Pre-dose (Day 1) and up to Day 8; Part A, FE and Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22; MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and B: AUC (0-inf): Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinite Time of EA1080 and its Metabolite | Part A and B, SAD: Pre-dose (Day 1) and up to Day 8; Part A, FE and Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22; MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and B: %AUCextrap: Percentage of AUC (0-inf) That is due to Extrapolation From tlast to Infinity of EA1080 and its Metabolite | SAD: Pre-dose (Day 1) and up to Day 8; FE and optional BA: Pre-dose (Day 1) and up to Day 15; MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and B: CL/F: Apparent Total Body Clearance of EA1080 and its Metabolite | Part A and B, SAD: Pre-dose (Day 1) and up to Day 8; Part A, FE and Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22; MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and B: Vz/F: Apparent Volume of Distribution During the Terminal Phase of EA1080 and its Metabolite | Part A and B, SAD: Pre-dose (Day 1) and up to Day 8; Part A, FE and Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22; MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and B: Ae: Amount of Drug EA1080 Excreted in Urine | Part A and B, SAD: Pre-dose (Day 1) and up to Day 5; Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 5; Part A and B, MAD: Pre-dose (Day 1) and up to Day 25 Part A and Day 21 for Part B
Parts A and B: fe: Percentage of EA1080 and its Metabolite Dose Excreted in Urine | Part A and B, SAD: Pre-dose (Day 1) and up to Day 5; Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 5; MAD: Pre-dose (Day 1) and up to Day 25 Part A and Day 21 for Part B
Parts A and B: CLR: Renal Clearance of EA1080 and its Metabolite | Part A and B, SAD: Pre-dose (Day 1) and up to Day 5; Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 5; MAD: Pre-dose (Day 1) and up to Day 25 Part A and Day 21 for Part B
Parts A and B: AUC (0-τ): Area Under the Plasma Concentration-time Curve From Time Zero to the Final Dosing Interval (τ) of EA1080 and its Metabolite | MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and Part B: Ctrough: Measured Plasma Concentration at the end of Each Dosing Interval of EA1080 and its Metabolite | MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and Part B: Cmax: Maximum Plasma Concentration Over the Dosing Period of EA1080 and its Metabolite | MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and Part B: AR(AUC): Accumulation Ratio For AUC0-τ of EA1080 and its Metabolite | MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and Part B: AR(Cmax): Accumulation Ratio For Cmax of EA1080 and its Metabolite | MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and Part B: AUC of EA1080 in Each Formulation | Part A and B, SAD: Pre-dose (Day 1) and up to Day 8; Part A, FE and Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22; MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and Part B: Cmax of EA1080 in Each Formulation | Part A and B, SAD: Pre-dose (Day 1) and up to Day 8; Part A, FE and Part B, SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22; MAD: Pre-dose (Day 1) and up to Day 28 Part A and up to Day 24 Part B
Parts A and Part B: AUC of EA1080 in Fed and Fasted State | Part A, FE: Pre-dose (Day 1) and up to Day 15; Part B SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22
Parts A and Part B: Cmax of EA1080 in Fed and Fasted State | Part A, FE: Pre-dose (Day 1) and up to Day 15; Part B SAD and additional FE: Pre-dose (Day 1) and up to Day 15; Part B, FE/BA: Pre-dose (Day 1) and up to Day 22

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond Pharmacology Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No